CLINICAL TRIAL: NCT02209584
Title: An Open Registry to Measure the Impact of Adding Genomic Testing (Prolaris®) on the Treatment Decision Following Biopsy in Newly Diagnosed Prostate Cancer Patients by Specialists
Brief Title: Open Registry Measuring Impact of Genomic Testing on Treatment Decision After Biopsy in Newly Diagnosed Prostate Cancer Patients
Acronym: PROCEDE-2000
Status: Completed | Type: Observational
Sponsor: Myriad Genetic Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PROCEDE-2000
Record Dates: First submitted 2014-04-29; First posted 2014-08-06 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2015-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
This registry is intended to measure the impact of Prolaris® testing on therapeutic decisions when added to standard clinical-pathological parameters in men with newly diagnosed prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed (≤6 months), untreated patients with histologically proven adenocarcinoma of the prostate that have the following characteristics.
* Clinically localized (no evidence on clinical or imaging studies of advanced disease.
* No hormonal therapy including LHRH agonist or antagonist, anti-androgen, 5-alpha reductase inhibitor, estrogens or exogenous androgens, when applicable.
* Sufficient amount of tissue remains from biopsy to perform genomic testing.

Exclusion Criteria:

* Patients with known history of hypogonadism will be excluded from the registry

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recently diagnosed treatment-naïve patients with early stage localized prostate cancer.
Sampling Method: Non-Probability Sample
Enrollment: 274 (Actual)
Dates: Start 2014-05; Primary Completion 2015-04-15 (Actual); Study Completion 2015-12-08 (Actual)

PRIMARY OUTCOMES:
Percentage change from the recorded PRE-Prolaris® test treatment option versus the ACTUAL treatment option of genomic risk assessment testing (Prolaris®). | 1 months

SECONDARY OUTCOMES:
Percentage change from the recorded PRE-Prolaris® test treatment option versus the POST-Prolaris® test treatment plan (prior to patient consultation). | 1 month

OTHER OUTCOMES:
Percentage change from the recorded PRE-Prolaris® test treatment option versus the POST-Prolaris® test treatment plan following consultation with the patient. | 1 month
The mean change in the physician's likelihood of recommending non-interventional therapy (watchful waiting or active surveillance) post-genomic testing compared to pre-genomic testing. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Richard Wenstrup, MD, Study Director — Myriad Genetic Laboratories, Inc.
Locations (1):
- University of Washington, Seattle, Washington, United States